CLINICAL TRIAL: NCT03662516
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL, 2-WAY CROSSOVER STUDY TO ESTIMATE THE EFFECT OF MULTIPLE DOSE PF-04965842 ON THE PHARMACOKINETICS OF SINGLE-DOSE ORAL CONTRACEPTIVE STEROIDS IN HEALTHY FEMALE SUBJECTS
Brief Title: A Study to Determine the Effects of PF-04965842 on the Pharmacokinetics of Oral Contraceptive Steroids in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B7451016
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Healthy Females
Keywords: PF-04965842
MeSH Terms: interventions — abrocitinib; Ethinyl Estradiol; Levonorgestrel; Contraceptives, Oral

STUDY DESIGN:
Intervention Model Description: Natural log transformed AUCinf, AUClast, and Cmax of EE and LN will be analyzed separately using a mixed effect model with sequence, period and treatment as fixed effects and subject within sequence as a random effect. Estimates of the adjusted mean differences (Test Reference) and corresponding 90% CIs will be obtained from the model. The adjusted mean differences and 90% CIs for the differences will be exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. OC (EE and LN) alone will be the Reference treatment, while the OC (EE and LN) coadministered with PF 04965842 will be the Test treatment.
  The absent of an effect of PF 04965842 on OC (EE and LN) will be concluded if the lower bound of 90% confidence interval for the ratio of adjusted geometric mean for AUCinf is ≥80%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Other): In Treatment Sequence 1, Period 1 Day 1, subjects will be dosed with a single administration of OC in the form of 1 PORTIA (EE and LN) or equivalent tablet, orally. OC (EE and LN) PK will then be assessed at pre dose and over 48 hours after OC dosing. Period 1 will be immediately followed by Period 2 with no washout. The 48 hours post-OC dose PK sample for Period 1 must be collected prior to receiving the first dose of PF 04965842 in Period 2. In Period 2, subjects will be dosed with 200 mg PF 04965842 PO QD for 9 days followed by administration of a single dose of OC oral tablet immediately after administration of a 200 mg dose of PF-04965842 on the morning of Day 10. OC PK in Period 2 will be assessed at pre dose and over 48 hours after OC dosing. Dosing with 200 mg PF 04965842 PO QD will continue until Day 11.
  Interventions: Drug: PF-04965842; Drug: Ethinyl estradiol (EE) and levonorgestrel (LN)
- Sequence 2 (Other): In Treatment Sequence 2, Period 1, subjects will be dosed with 200 mg PF 04965842 PO QD for 9 days followed by administration of a single dose of OC oral tablet immediately after administration of a 200 mg dose of PF-04965842 on the morning of Day 10. OC PK will be assessed at pre dose and over 48 hours following OC dosing. Dosing with 200 mg PF 04965842 PO QD will continue until Day 11. Subjects will then undergo a washout period of at least 10 days (Day -1 of Period 2 starts 10 days after Day 12 of Period 1). In Period 2 subjects will be dosed with a single OC administration on Day 1. OC PK will then be assessed at pre dose and over 48 hours after OC dose.
  Interventions: Drug: PF-04965842; Drug: Ethinyl estradiol (EE) and levonorgestrel (LN)

INTERVENTIONS:
Drug: PF-04965842 — Orally bioavailable small molecule that selectively inhibits JAK 1 by blocking the adenosine triphosphate (ATP) binding site.
  Other Names: JAK 1 inhibitor
Drug: Ethinyl estradiol (EE) and levonorgestrel (LN) — Single dose of Oral tablet containing 30 ug EE and 150 ug of LN
  Other Names: Oral contraceptive

SUMMARY:
This is a Phase 1, randomized, 2 way crossover, open-label study of the effect of multiple-dose PF 04965842 on single-dose OC PK in healthy female subjects. Subjects will be randomized to 1 of 2 treatment sequences. A total of 16 healthy female subjects (8 in each treatment sequence) will be enrolled in the study. Each treatment sequence will consist of 2 periods.

DETAILED DESCRIPTION:
In Treatment Sequence 1, Period 1 Day 1, subjects will be dosed with a single administration of OC in the form of 1 PORTIA (ethyinyl estradiol [EE] and levonorgestrel [LN]) or equivalent tablet, orally. OC (EE and LN) PK will then be assessed at pre dose and over 48 hours after OC dosing. Period 1 will be immediately followed by Period 2 with no washout. The 48 hours post-OC dose PK sample for Period 1 must be collected prior to receiving the first dose of PF 04965842 in Period 2. In Period 2, subjects will be dosed with 200 mg PF 04965842 PO QD for 9 days followed by administration of a single dose of OC oral tablet immediately after administration of a 200 mg dose of PF-04965842 on the morning of Day 10. OC PK in Period 2 will be assessed at pre dose and over 48 hours after OC dosing. Dosing with 200 mg PF 04965842 PO QD will continue until Day 11.

In Treatment Sequence 2, Period 1, subjects will be dosed with 200 mg PF 04965842 PO QD for 9 days followed by administration of a single dose of OC oral tablet immediately after administration of a 200 mg dose of PF-04965842 on the morning of Day 10. OC PK will be assessed at pre dose and over 48 hours following OC dosing. Dosing with 200 mg PF 04965842 PO QD will continue until Day 11. Subjects will then undergo a washout period of at least 10 days (Day -1 of Period 2 starts 10 days after Day 12 of Period 1). In Period 2 subjects will be dosed with a single OC administration on Day 1. OC PK will then be assessed at pre dose and over 48 hours after OC dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of both childbearing and non-childbearing potential who, at the time of Screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure (BP) and pulse rate measurement, 12 lead ECG, or clinical laboratory tests.

Female subjects of non-childbearing potential must meet at least 1 of the following criteria:

1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state;
2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
3. Have medically confirmed ovarian failure. All other female subjects (including female subjects with tubal ligations) are considered to be of childbearing potential.

   * Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
   * Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
   * Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, gynecologic or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Evidence of acute exacerbation of dermatological condition (eg, AD or psoriasis) or visible rash present during physical examination.
* Subjects, who according to the product label for OC, would be at increased risk if dosed with OC.

Based on PORTIA product label, combination OCs should not be used in women with any of the following conditions:

1. Thrombophlebitis or thromboembolic disorders.
2. A past history of deep-vein thrombophlebitis or thromboembolic disorders.
3. Cerebral-vascular or coronary artery disease.
4. Thrombogenic valvulopathies.
5. Thrombogenic rhythm disorders.
6. Diabetes mellitus with vascular involvement.
7. Uncontrolled hypertension.
8. Known or suspected carcinoma of the breast.
9. Carcinoma of the endometrium or other known or suspected estrogen-dependent neoplasia.
10. Undiagnosed abnormal genital bleeding.
11. Cholestatic jaundice of pregnancy or jaundice with prior pill use.
12. Hepatic adenomas or carcinomas, or active liver disease, as long as liver function has not returned to normal.
13. Known or suspected pregnancy.
14. Hypersensitivity to any of the components of Portia (LN and EE tablets).
15. Are receiving Hepatitis C drug combinations containing ombitasvir/paritaprevir/ritonavir, with or without dasabuvir, due to the potential for alanine aminotransferase (ALT) elevations.

    * Any condition possibly affecting drug absorption (eg, gastrectomy).
    * A positive urine drug test.
    * History of regular alcohol consumption exceeding 7 drinks/week for female subjects (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months before Screening.
    * Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product (whichever is longer).
    * Screening supine systolic BP <90 mm Hg or 140 mm Hg following at least 5 minutes of supine rest or Screening supine diastolic BP <50 mm Hg or 90 mm Hg following at least 5 minutes of supine rest.

If a subject meets any of these criteria, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the subject's eligibility.

* Screening supine 12 lead ECG demonstrating a corrected QT (QTc) interval >450 msec or a QRS interval >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the subject's eligibility.
* Subjects with ANY of the following abnormalities in clinical laboratory tests at Screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

  * Aspartate aminotransferase (AST) or ALT level >= 1.5 × upper limit of normal (ULN);
  * Total bilirubin (TBili) level > 1 × ULN;
* Use of CYP2C19 inhibitors (eg, fluconazole, fluoxetine, fluvoxamine, ticlopidine omeprazole, voriconazole, cimetidine, esomeprazole, and felbamate) or inducers (eg, rifampin, ritonavir, efavirenz, enzalutamide, phenytoin, and St. John's Wort) within 28 days or 5 half-lives (whichever is longer) prior to dosing.
* Use of CYP2C9 inhibitors (eg, amiodarone, felbamate, fluconazole, miconazole, piperine, diosmin, disulfiram, fluvastatin, fluvoxamine, voriconazole, efavirenz, isoniazid) or inducers (eg, aprepitant, carbamazepine, enzalutamide, rifampin, ritonavir, nevirapine, phenobarbital, and St. John's Wort) within 28 days or 5 half-lives (whichever is longer) prior to dosing.
* Use of CYP3A4 inhibitors (eg, ketoconazole, ciprofloxacin, diltiazem) or other inducers (eg, phenytoin, carbamazepine) within 28 days or 5 half-lives (whichever is longer) prior to dosing.
* Known relevant history of elevated liver function tests (LFTs).
* History of active or latent or inadequately treated tuberculosis (TB) infection, or a positive QuantiFERON-TB Gold test.
* Any history of chronic infections, any history of recurrent infections, any history of latent infections, or any acute infection within 2 weeks of Screening.

  * History of disseminated herpes zoster, or disseminated herpes simplex, or recurrent localized dermatomal herpes zoster.
  * History of systemic infection requiring hospitalization, parenteral antimicrobial therapy, or considered clinically significant by the investigator within 6 months prior to Screening.
* History of receiving a live vaccine within 6 weeks prior to the first dose of investigational product, or is expected to receive a live vaccine within 6 weeks after the last dose of investigational product.
* Have a known immunodeficiency disorder or a first-degree relative with a hereditary immunodeficiency.
* History or evidence of any malignancies with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin, or cervical carcinoma in situ.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of investigational product. As an exception, acetaminophen/paracetamol may be used at doses of <= 1 g/day. Limited use of nonprescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case by case basis following approval by the sponsor.

Herbal supplements and hormonal methods of contraception (including oral and transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone releasing intrauterine devices [IUDs], vaginal ring, and postcoital contraceptive methods) and hormone replacement therapy must have been discontinued at least 28 days prior to the first dose of investigational product.

Use of hormone based intravaginal creams (i.e., Estrace) for treatment of vaginal dryness, itching, or burning due to menopause and/or vulvovaginal atrophy Depo Provera must have been discontinued at least 6 months prior to the first dose of investigational product.

* Use of tobacco- or nicotine-containing products within 3 months of Screening or a positive urine cotinine at Screening.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb).

A positive hepatitis B surface antibody (HepBsAb) finding as a result of subject vaccination is permissible.

* A current or past medical history of conditions associated with thrombocytopenia, coagulopathy, or platelet dysfunction.
* Unwilling or unable to comply with the criteria in the Lifestyle Requirements section of this protocol.
* Unwillingness to use an additional form of contraception for the duration of the study and for the specified time after follow-up.
* History of discontinued use of OCs for medical reasons.
* Pregnant female subjects; breastfeeding female subjects; females of childbearing potential who do not agree to use an acceptable method of nonhormonal contraception.
* Subjects who are investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy female subjects of both childbearing and non-childbearing potential.
Enrollment: 17 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-01-19 (Actual); Study Completion 2019-01-19 (Actual)

PRIMARY OUTCOMES:
AUCinf for EE | 0 (pre-dose),1, 1.5. 2, 4, 6, 8, 12, 24 and 48 hours post-dose.
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
AUCinf for LN | 0 (pre-dose), 1, 1.5, 2, 4, 6, 8, 12, 24 and 48 hours post-dose.
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).

SECONDARY OUTCOMES:
Laboratory tests | Baseline through study completion, approximately 15 days for sequence 1 and 25 days for sequence 2.
  Number of subjects with laboratory test abnormalities.
Adverse Events (AEs) | Baseline (Day 0) up to 28 days after last dose of study drug
  Number of subjects with treatment-related treatment emergent adverse events.
Vital signs | Baseline through study completion, approximately 15 days for sequence 1 and 25 days for sequence 2.
  Number of subjects with vital sign data (blood pressure, pulse rate, and oral temperature) of potential clinical concern.
12-lead ECGs | Day 1 and Day 12 of PF-04965842 and OC co-administration period.
  Number of subjects with ECG data of potential clinical concern.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Wang X, Dowty ME, Tripathy S, Le VH, Huh Y, Curto M, Winton JA, O'Gorman MT, Chan G, Malhotra BK. Assessment of the Effects of Abrocitinib on the Pharmacokinetics of Probe Substrates of Cytochrome P450 1A2, 2B6 and 2C19 Enzymes and Hormonal Oral Contraceptives in Healthy Individuals. Eur J Drug Metab Pharmacokinet. 2024 May;49(3):367-381. doi: 10.1007/s13318-024-00893-5. Epub 2024 Mar 30. PMID 38554232
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451016